CLINICAL TRIAL: NCT07290114
Title: Mesh-Free Versus Mesh-Based Surgery for Female Stress Urinary Incontinence: A Prospective Comparison of Pubo-Urethral Ligament Plication and Transobturator Tape With Short-Term Patient-Centered Outcomes
Brief Title: Mesh-Free Versus Mesh-Based Surgery for Female Stress Urinary Incontinence: A Prospective Comparison of Pubo-Urethral Ligament Plication and Transobturator Tape
Acronym: PLP-TOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mehmet Incebıyik (Other)
Responsible Party: Sponsor-Investigator, Mehmet Incebıyik, Assistant Professor of Obstetrics and Gynecology, Harran University
Organization: Harran University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HU-SUI-PLP-TOT-2025
Record Dates: First submitted 2025-12-04; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Stress Urinary Incontinence (SUI)
Keywords: Stress Urinary Incontinence, Pubo-Urethral Ligament Plication, PLP, Transobturator Tape, TOT, Mesh-free surgery, Midurethral sling
MeSH Terms: conditions — Urinary Incontinence, Stress; Pelizaeus-Merzbacher Disease | interventions — Suburethral Slings

STUDY DESIGN:
Intervention Model Description: Two-arm prospective parallel comparison of mesh-free PLP versus mesh-based TOT surgical techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLP Arm (Experimental): Patients undergoing mesh-free Pubo-Urethral Ligament Plication (PLP), a native tissue surgical technique performed to reinforce urethral support without the use of synthetic mesh.
  Interventions: Procedure: Pubo-Urethral Ligament Plication (PLP)
- TOT Arm (Active Comparator): Patients undergoing the Transobturator Tape (TOT) procedure, a widely used mesh-based midurethral sling technique performed to provide urethral support via the transobturator route.
  Interventions: Procedure: Transobturator Tape (TOT)

INTERVENTIONS:
Procedure: Pubo-Urethral Ligament Plication (PLP) — A mesh-free native tissue surgical technique that reinforces urethral support by plicating the pubo-urethral ligament. The procedure aims to restore midurethral stability without the use of synthetic mesh.
  Arms: PLP Arm
Procedure: Transobturator Tape (TOT) — A mesh-based midurethral sling procedure performed through the transobturator route to provide urethral support. The tape is positioned under the midurethra to treat stress urinary incontinence.
  Arms: TOT Arm

SUMMARY:
This prospective clinical study aims to compare the short-term effectiveness, safety, and patient-reported outcomes of two surgical techniques used for the treatment of female stress urinary incontinence (SUI): Pubo-Urethral Ligament Plication (PLP), a mesh-free native tissue repair method, and the Transobturator Tape (TOT) procedure, a commonly used mesh-based mid-urethral sling technique. The study evaluates continence improvement, perioperative and postoperative complications, operative time, hospital stay, postoperative pain, and patient satisfaction. The goal is to provide evidence on whether a mesh-free surgical option such as PLP can offer comparable outcomes to mesh-based TOT, particularly for patients seeking alternatives to synthetic materials.

DETAILED DESCRIPTION:
This is a single-center, prospective, comparative clinical study evaluating two established surgical interventions for female stress urinary incontinence (SUI): Pubo-Urethral Ligament Plication (PLP) and Transobturator Tape (TOT). PLP is a mesh-free native tissue repair technique that reinforces pubo-urethral support by plicating the periurethral tissues. TOT, a mesh-based mid-urethral sling procedure, provides support to the urethra through the placement of a synthetic tape via the transobturator route.

Eligible patients with a clinical diagnosis of SUI who elect to undergo surgical treatment will be allocated to one of the two interventions based on shared decision-making between the surgeon and the patient. The study will collect demographic data, operative parameters, perioperative complications, and short-term postoperative outcomes. Continence outcomes will be assessed using validated questionnaires such as the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF), as well as objective clinical evaluation during follow-up visits. Pain levels, urinary retention, de-novo urgency, wound complications, and overall patient satisfaction will also be recorded.

The primary aim of the study is to compare early continence improvement between the PLP and TOT procedures. Secondary aims include comparing perioperative and postoperative complications, operative time, postoperative pain, hospital discharge time, and patient-reported satisfaction. By directly comparing a mesh-free native tissue technique with a commonly used mesh-based sling, this study seeks to provide updated, patient-centered data that may guide surgical decision-making, especially in settings where mesh-related concerns or patient preference favor native tissue repair options.

ELIGIBILITY:
Inclusion Criteria:

Female patients aged 18-80 years

Clinical diagnosis of stress urinary incontinence

Failure of conservative management (pelvic floor exercises or medical therapy)

Desire to undergo surgical treatment (PLP or TOT)

Ability to provide informed consent

Willingness to attend postoperative follow-up visits

Exclusion Criteria:

* Mixed urinary incontinence with predominant urge symptoms

Active urinary tract infection

Pelvic organ prolapse ≥ stage II

Previous anti-incontinence surgery

Neurological diseases affecting bladder function

Pregnancy or planning pregnancy during follow-up

Uncontrolled diabetes, bleeding disorders, or contraindications to surgery

Use of medications affecting bladder function (e.g., anticholinergics)

Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Improvement in Stress Urinary Incontinence Symptoms (ICIQ-SF Score) | 6-24 weeks postoperatively
  Change in the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) score from baseline to postoperative 6 weeks. Lower scores indicate improvement in symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: MEHMET İNCEBIYIK, MD, Principal Investigator — Harran University
Locations (1):
- Harran University Research and Application Hospital, Şanliurfa, HALİLİYE, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided